CLINICAL TRIAL: NCT01394978
Title: AirTight: A Prospective Controlled Post-Approval Study of NeoMend ProGEL™ Pleural Air Leak Sealant in the Treatment of Visible Pleural Air Leaks After Standard Pleural Closure
Brief Title: NeoMend ProGEL™ Pleural Air Leak Sealant Post-Approval Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEO09-100
Record Dates: First submitted 2011-07-13; First posted 2011-07-15 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Lung Cancer; Lung Tumor
Keywords: Pleural air leak; Pulmonary resection; Open thoracotomy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Other): No treatment.
  Interventions: Other: Control
- ProGEL Pleural Air Leak Sealant with standard surgical closure (Experimental): Standard surgical closure (suturing or stapling of visible air leaks incurred during resection of lung parenchyma) plus Progel Pleural Air Leak Sealant.
  Interventions: Device: ProGEL Pleural Air Leak Sealant with standard surgical closure
- ProGEL Pleural Air Leak Sealant without standard surgical closure (Experimental): Progel Pleural Air Leak Sealant without standard surgical closure (without suturing or stapling of visible air leaks incurred during resection of lung parenchyma).
  Interventions: Device: ProGEL Pleural Air Leak Sealant without standard surgical closure

INTERVENTIONS:
Other: Control — Standard surgical techniques including staples and sutures.
  Arms: Control
Device: ProGEL Pleural Air Leak Sealant with standard surgical closure — ProGEL is a single-use medical device that is formed as a result of mixing two components: (1) a solution of human serum albumin (HSA) and (2) a synthetic cross-linking component of polyethylene glycol (PEG). Standard closure means, for example, suturing or stapling of visible air leaks incurred during resection of lung parenchyma.
  Arms: ProGEL Pleural Air Leak Sealant with standard surgical closure
Device: ProGEL Pleural Air Leak Sealant without standard surgical closure — ProGEL is a single-use medical device that is formed as a result of mixing two components: (1) a solution of human serum albumin (HSA) and (2) a synthetic cross-linking component of polyethylene glycol (PEG). Standard closure means, for example, suturing or stapling of visible air leaks incurred during resection of lung parenchyma.
  Arms: ProGEL Pleural Air Leak Sealant without standard surgical closure

SUMMARY:
The purpose of this post approval study is to further characterize the safety profile of the ProGEL™ Pleural Air Leak Sealant in commercial use, with specific reference to long-term safety over 90 days of follow-up.

DETAILED DESCRIPTION:
Patients having open thoracotomy involving lung resection surgery will be considered for the study. Subjects will be examined for adverse events and complications from either the treatment or the procedure. Follow-up visits are required at 30 days and 90 days after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for an open thoracotomy for lung resection
* Has at least one or more intraoperative visible air leak >= 2 mm following the lung resection surgery

Exclusion Criteria:

* Pregnant or breast feeding
* History of an allergic reaction to Human Serum Albumin
* Has a significant clinical disease or condition
* Had previous open thoracotomy procedures
* Unable to participate in all necessary study activities due to physical or mental limitations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2011-06; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Cerfolio, MD, Principal Investigator — University of Alabama in Birmingham; Daniel L. Miller, MD, Principal Investigator — WellStar Research Institute
Locations (18):
- United States (18):
  - St. Vincent Birmingham & St. Vincent East, Birmingham, Alabama
  - University of Alabama in Birmingham, Birmingham, Alabama
  - Jacksonville Center for Research, Jacksonville, Florida
  - Moffit Cancer Center, Tampa, Florida
  - WellStar Research Institute, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - St. Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Mass General Hospital, Boston, Massachusetts
  - Brigham Womens' Hospital, Boston, Massachusetts
  - Beth Israel Deconess Medical Center, Boston, Massachusetts
  - UMass Memorial Medical, Worcester, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - Dean Foundation for Health, Research and Education, Inc., Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The original Protocol was designed to study ProGel (any usage) versus no ProGel. After the study was completed, the FDA requested that the ProGel group be broken out by patients with standard closure, and without.
Groups:
- ProGEL Pleural Air Leak Sealant: Standard surgical technique plus Progel Pleural Air Leak Sealant.
  ProGEL Pleural Air Leak Sealant: ProGEL is a single-use medical device that is formed as a result of mixing two components: (1) a solution of human serum albumin (HSA) and (2) a synthetic cross-linking component of polyethylene glycol (PEG).
Period: Overall Study
Arm/Group | Control | ProGEL Pleural Air Leak Sealant
Started | 168 | 276
Completed | 147 | 245
Not Completed | 21 | 31
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Lost to Follow-up | 13 | 20
Not completed — Death | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- ProGEL Pleural Air Leak Sealant With Standard Surgical Closure: ProGEL Pleural Air Leak Sealant: ProGEL is a single-use medical device that is formed as a result of mixing two components: (1) a solution of human serum albumin (HSA) and (2) a synthetic cross-linking component of polyethylene glycol (PEG).
  Standard closure, for example, by suturing or stapling, of visible air leaks incurred during resection of lung parenchyma.
- ProGEL Pleural Air Leak Sealant Without Standard Surgical Closure: ProGEL Pleural Air Leak Sealant: ProGEL is a single-use medical device that is formed as a result of mixing two components: (1) a solution of human serum albumin (HSA) and (2) a synthetic cross-linking component of polyethylene glycol (PEG).
  Without standard closure, for example, suturing or stapling, of visible air leaks incurred during resection of lung parenchyma.
- Total: Total of all reporting groups
Arm/Group | Control | ProGEL Pleural Air Leak Sealant With Standard Surgical Closure | ProGEL Pleural Air Leak Sealant Without Standard Surgical Closure | Total
Number analyzed (Participants) | 168 | 169 | 107 | 444
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 69 | 78 | 44 | 191
  >=65 years | 99 | 91 | 63 | 253
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (11.46) | 64.8 (11.30) | 66.7 (9.10) | 65.6 (10.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 81 | 55 | 217
  Male | 87 | 88 | 52 | 227
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 156 | 161 | 97 | 414
  Race/Ethnicity: Black | 8 | 8 | 7 | 23
  Race/Ethnicity: Asian | 1 | 0 | 1 | 2
  Race/Ethnicity: Hispanic | 2 | 0 | 1 | 3
  Race/Ethnicity: Other | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 168 | 169 | 107 | 444
Height [Mean (Standard Deviation); unit: centimeters] | 169.3 (9.93) | 171.0 (9.72) | 168.6 (9.40) | 169.8 (9.74)
Weight [Mean (Standard Deviation); unit: kilograms] | 79.9 (19.75) | 82.0 (21.43) | 78.0 (18.48) | 80.3 (20.22)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.8 (6.16) | 27.9 (6.52) | 27.3 (5.47) | 27.7 (6.11)

OUTCOME MEASURES:

1. Primary Outcome: Safety Endpoints
Description: * Pulmonary adverse events: pneumothorax, persistent air leak, late onset air leak, residual pleural space, and acute respiratory distress syndrome
  * Renal adverse events
  * Cardiac adverse events
  * Death (all causes)
  * Hospital readmission
Time Frame: 90 days
Population: Units analyzed represents the number of adverse events that occurred among all study participants in each arm.
  Also, the original Protocol was designed to study ProGel (any usage) versus no ProGel. After the study was completed, the FDA requested that the ProGel group be broken out by patients with standard closure, and without.
Measure: Count of Units; unit: Events
Units Other Than Participants: Events
Arm/Group | Control | ProGEL Pleural Air Leak Sealant
Number analyzed (Participants) | 168 | 276
Number analyzed (Events) | 111 | 191
Events
  Pneumothorax | 22 | 48
  Persistent air leak | 25 | 40
  Late onset air leak | 1 | 6
  Residual pleural space | 1 | 1
  Acute respiratory distress syndrome | 1 | 3
  Renal abnormalities | 5 | 7
  Myocardial Infarction | 0 | 2
  Atrial Arrythmia | 29 | 48
  Ventricular Arrythmia | 5 | 4
  Cardiac Arrest, Resuscitated | 0 | 2
  Death, all causes | 6 | 7
  Hospital readmission | 16 | 23

ADVERSE EVENTS:
Time Frame: 90 days post-index procedure
Groups:
- ProGEL Pleural Air Leak Sealant With Standard Surgical Closure: ProGEL Pleural Air Leak Sealant: ProGEL is a single-use medical device that is formed as a result of mixing two components: (1) a solution of human serum albumin (HSA) and (2) a synthetic cross-linking component of polyethylene glycol (PEG).
  Standard surgical closure (standard closure with, sutures or staples, for example) plus Progel Pleural Air Leak Sealant.
- ProGEL Pleural Air Leak Sealant Without Standard Surgical Closure: ProGEL Pleural Air Leak Sealant: ProGEL is a single-use medical device that is formed as a result of mixing two components: (1) a solution of human serum albumin (HSA) and (2) a synthetic cross-linking component of polyethylene glycol (PEG).
  Progel Pleural Air Leak Sealant without standard surgical closure (standard closure with, sutures or staples, for example).
Arm/Group | Control | ProGEL Pleural Air Leak Sealant With Standard Surgical Closure | ProGEL Pleural Air Leak Sealant Without Standard Surgical Closure
All-Cause Mortality (participants affected / at risk) | 6/168 | 5/169 | 2/107
Serious Adverse Events (participants affected / at risk) | 40/168 | 37/169 | 27/107
Other Adverse Events (participants affected / at risk) | 39/168 | 52/169 | 33/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=168) | ProGEL Pleural Air Leak Sealant With Standard Surgical Closure (N=169) | ProGEL Pleural Air Leak Sealant Without Standard Surgical Closure (N=107)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 8 | 10 | 8
Persistent air leak (Respiratory, thoracic and mediastinal disorders) | 15 | 18 | 5
Late onset air leak (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4
Residual Plueral Space (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Renal abnormalities (Renal and urinary disorders) | 2 | 3 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 1 | 1
Atrial Arrhythmia (Cardiac disorders) | 6 | 1 | 1
Ventricular Arrythmia (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest, resuscitated (Cardiac disorders) | 0 | 1 | 1
Death, All Causes (General disorders) | 6 | 5 | 2
Hospital Readmission (General disorders) | 14 | 8 | 12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=168) | ProGEL Pleural Air Leak Sealant With Standard Surgical Closure (N=169) | ProGEL Pleural Air Leak Sealant Without Standard Surgical Closure (N=107)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 22 (22) | 11 (11)
Persistent Air Leak (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 11 (22) | 7 (11)
Atrial Arrhythmia (Cardiac disorders) | 20 (20) | 26 (26) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No